CLINICAL TRIAL: NCT02392182
Title: Understanding the Lung Microbiome in HIV-Infected & HIV-Uninfected Individuals
Brief Title: Lung HIV Microbiome Project (Michigan Site)
Acronym: LHMP
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jeffrey L. Curtis, Professor of Internal Medicine, University of Michigan
Other Study IDs: Curtis 0036
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Healthy Participants; Tobacco Use Disorder; Human Microbiome
Keywords: lung
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Oral rinse Nasal swap Bronchoalveolar lavage
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- healthy volunteers: no intervention to be administered in this observational study, although all participants will undergo fiberoptic bronchoscopy.
  Interventions: Other: Fiberoptic bronchoscopy

INTERVENTIONS:
Other: Fiberoptic bronchoscopy — All subjects will undergo a research fiberoptic bronchoscopy under moderate conscious sedation. There is no randomization

SUMMARY:
In its original phase, this cohort study recruited subjects who were either HIV-positive or HIV-negative healthy controls, to analyze the community structure of the lung microbiome. Original recruitment was planned to occur both at the University of Michigan Medical Center and clinics, and at VA Ann Arbor Healthcare System.

Enrollment for the original cohort is completed, and all current activity of this project is occurring at VA Ann Arbor, where both Veteran subjects and non-Veteran subjects are eligible to participate. This study is currently recruiting only healthy HIV-negative subjects. Participation, described below, involves a research bronchoscopy procedure.

DETAILED DESCRIPTION:
This is a non-interventional cohort study with single time point cross-sectional comparisons and longitudinal analyses, with the primary study aims of: evaluating how the immune deficiency associated with HIV infection influences the lung microbiome and lung function, and evaluating changes in lung microbiota over time. The study also aims to characterize the microbiome of the lower respiratory tract, determine the relationship between the lower respiratory Microbiome and the upper respiratory and gastrointestinal tract microbiomes, evaluate the influence of smoking on the microbiome compared with the influence of smoking on pulmonary function and respiratory systems, and to evaluate how Pneumocystis infection influences HIV-infected and HIV-uninfected individuals.

ELIGIBILITY:
Inclusion Criteria:

* Negative HIV testing (by ELISA) during initial study visit
* No signs of respiratory infection at enrollment, such as: fever; recent change in quantity of quality of sputum; chest pain; recent change in shortness of breath or exertional activity
* Willing and able to sign the informed consent document
* If female of child-bearing potential, negative pregnancy test during initial study visit

Exclusion Criteria:

* Pregnancy
* Signs or symptoms of respiratory infection at enrollment
* Unwilling or unable to sign the informed consent document
* Unstable heart disease
* Other systemic disease and unlikely to survive at least 2 years
* Mental incompetence
* Participation in another interventional protocol within the last 6 weeks
* Use of antibiotics for a lung infection within the last 4 weeks
* Renal Failure (creatinine >3)
* Child's Class C Cirrhosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals with no more than mild treated chronic diseases that would not preclude a research bronchoscopy under moderate conscious sedation. Both never-smokers and active smokers are welcome.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2009-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Lung bacterial microbiome community structure | at time of bronchoscopy
  biological samples will be analyzed by culture-independent microbiological and bioinformatic techniques to determine the constituent members of the bacterial microbiome at each sampled site, to the level of "operational taxonomic unit" at 97% similarity to published sequences.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L. Curtis, MD, Principal Investigator — Professor of Internal Medicine & Staff Physician, VA Ann Arbor
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
deidentified data and biological specimens deposited with NIH BioLNCC

REFERENCES:
- [Background] Twigg HL 3rd, Morris A, Ghedin E, Curtis JL, Huffnagle GB, Crothers K, Campbell TB, Flores SC, Fontenot AP, Beck JM, Huang L, Lynch S, Knox KS, Weinstock G; Lung HIV Microbiome Project. Use of bronchoalveolar lavage to assess the respiratory microbiome: signal in the noise. Lancet Respir Med. 2013 Jul;1(5):354-6. doi: 10.1016/S2213-2600(13)70117-6. Epub 2013 Jul 8. No abstract available. PMID 24429191
- [Background] Dickson RP, Erb-Downward JR, Huffnagle GB. The role of the bacterial microbiome in lung disease. Expert Rev Respir Med. 2013 Jun;7(3):245-57. doi: 10.1586/ers.13.24. PMID 23734647
- [Background] Dickson RP, Erb-Downward JR, Freeman CM, Walker N, Scales BS, Beck JM, Martinez FJ, Curtis JL, Lama VN, Huffnagle GB. Changes in the lung microbiome following lung transplantation include the emergence of two distinct Pseudomonas species with distinct clinical associations. PLoS One. 2014 May 15;9(5):e97214. doi: 10.1371/journal.pone.0097214. eCollection 2014. PMID 24831685
- [Background] Dickson RP, Erb-Downward JR, Huffnagle GB. Towards an ecology of the lung: new conceptual models of pulmonary microbiology and pneumonia pathogenesis. Lancet Respir Med. 2014 Mar;2(3):238-46. doi: 10.1016/S2213-2600(14)70028-1. PMID 24621685
- [Background] Dickson RP, Martinez FJ, Huffnagle GB. The role of the microbiome in exacerbations of chronic lung diseases. Lancet. 2014 Aug 23;384(9944):691-702. doi: 10.1016/S0140-6736(14)61136-3. PMID 25152271
- [Background] Scales BS, Dickson RP, LiPuma JJ, Huffnagle GB. Microbiology, genomics, and clinical significance of the Pseudomonas fluorescens species complex, an unappreciated colonizer of humans. Clin Microbiol Rev. 2014 Oct;27(4):927-48. doi: 10.1128/CMR.00044-14. PMID 25278578
- [Background] Dickson RP, Erb-Downward JR, Prescott HC, Martinez FJ, Curtis JL, Lama VN, Huffnagle GB. Intraalveolar Catecholamines and the Human Lung Microbiome. Am J Respir Crit Care Med. 2015 Jul 15;192(2):257-9. doi: 10.1164/rccm.201502-0326LE. No abstract available. PMID 26177175
- [Background] Curtis JL, Freeman CM, Huffnagle GB. "B" for Bad, Beneficial, or Both? Lung Lymphoid Neogenesis in Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2015 Sep 15;192(6):648-51. doi: 10.1164/rccm.201506-1230ED. No abstract available. PMID 26371807
- [Background] Curtis JL, Freeman CM. Why do we need a nonhuman primate model of smoking-induced COPD? Am J Pathol. 2015 Mar;185(3):610-3. doi: 10.1016/j.ajpath.2014.12.002. Epub 2015 Jan 7. PMID 25576784
- [Background] Huang YJ, Erb-Downward JR, Dickson RP, Curtis JL, Huffnagle GB, Han MK. Understanding the role of the microbiome in chronic obstructive pulmonary disease: principles, challenges, and future directions. Transl Res. 2017 Jan;179:71-83. doi: 10.1016/j.trsl.2016.06.007. Epub 2016 Jun 23. PMID 27392936
- [Background] Adar SD, Huffnagle GB, Curtis JL. The respiratory microbiome: an underappreciated player in the human response to inhaled pollutants? Ann Epidemiol. 2016 May;26(5):355-9. doi: 10.1016/j.annepidem.2016.03.010. Epub 2016 Apr 7. PMID 27161078
- [Result] Lozupone C, Cota-Gomez A, Palmer BE, Linderman DJ, Charlson ES, Sodergren E, Mitreva M, Abubucker S, Martin J, Yao G, Campbell TB, Flores SC, Ackerman G, Stombaugh J, Ursell L, Beck JM, Curtis JL, Young VB, Lynch SV, Huang L, Weinstock GM, Knox KS, Twigg H, Morris A, Ghedin E, Bushman FD, Collman RG, Knight R, Fontenot AP; Lung HIV Microbiome Project. Widespread colonization of the lung by Tropheryma whipplei in HIV infection. Am J Respir Crit Care Med. 2013 May 15;187(10):1110-7. doi: 10.1164/rccm.201211-2145OC. PMID 23392441
- [Result] Morris A, Beck JM, Schloss PD, Campbell TB, Crothers K, Curtis JL, Flores SC, Fontenot AP, Ghedin E, Huang L, Jablonski K, Kleerup E, Lynch SV, Sodergren E, Twigg H, Young VB, Bassis CM, Venkataraman A, Schmidt TM, Weinstock GM; Lung HIV Microbiome Project. Comparison of the respiratory microbiome in healthy nonsmokers and smokers. Am J Respir Crit Care Med. 2013 May 15;187(10):1067-75. doi: 10.1164/rccm.201210-1913OC. PMID 23491408
- [Result] Beck JM, Schloss PD, Venkataraman A, Twigg H 3rd, Jablonski KA, Bushman FD, Campbell TB, Charlson ES, Collman RG, Crothers K, Curtis JL, Drews KL, Flores SC, Fontenot AP, Foulkes MA, Frank I, Ghedin E, Huang L, Lynch SV, Morris A, Palmer BE, Schmidt TM, Sodergren E, Weinstock GM, Young VB; Lung HIV Microbiome Project. Multicenter Comparison of Lung and Oral Microbiomes of HIV-infected and HIV-uninfected Individuals. Am J Respir Crit Care Med. 2015 Dec 1;192(11):1335-44. doi: 10.1164/rccm.201501-0128OC. PMID 26247840
- [Result] Erb-Downward JR, Sadighi Akha AA, Wang J, Shen N, He B, Martinez FJ, Gyetko MR, Curtis JL, Huffnagle GB. Use of direct gradient analysis to uncover biological hypotheses in 16s survey data and beyond. Sci Rep. 2012;2:774. doi: 10.1038/srep00774. Epub 2012 Oct 26. PMID 23336065
- [Result] Dickson RP, Erb-Downward JR, Prescott HC, Martinez FJ, Curtis JL, Lama VN, Huffnagle GB. Cell-associated bacteria in the human lung microbiome. Microbiome. 2014 Aug 18;2:28. doi: 10.1186/2049-2618-2-28. eCollection 2014. PMID 25206976
- [Result] Venkataraman A, Bassis CM, Beck JM, Young VB, Curtis JL, Huffnagle GB, Schmidt TM. Application of a neutral community model to assess structuring of the human lung microbiome. mBio. 2015 Jan 20;6(1):e02284-14. doi: 10.1128/mBio.02284-14. PMID 25604788
- [Result] Bassis CM, Erb-Downward JR, Dickson RP, Freeman CM, Schmidt TM, Young VB, Beck JM, Curtis JL, Huffnagle GB. Analysis of the upper respiratory tract microbiotas as the source of the lung and gastric microbiotas in healthy individuals. mBio. 2015 Mar 3;6(2):e00037. doi: 10.1128/mBio.00037-15. PMID 25736890
- [Result] Dickson RP, Erb-Downward JR, Freeman CM, McCloskey L, Beck JM, Huffnagle GB, Curtis JL. Spatial Variation in the Healthy Human Lung Microbiome and the Adapted Island Model of Lung Biogeography. Ann Am Thorac Soc. 2015 Jun;12(6):821-30. doi: 10.1513/AnnalsATS.201501-029OC. PMID 25803243
- [Result] Erb-Downward JR, Thompson DL, Han MK, Freeman CM, McCloskey L, Schmidt LA, Young VB, Toews GB, Curtis JL, Sundaram B, Martinez FJ, Huffnagle GB. Analysis of the lung microbiome in the "healthy" smoker and in COPD. PLoS One. 2011 Feb 22;6(2):e16384. doi: 10.1371/journal.pone.0016384. PMID 21364979
- [Result] Qin S, Clausen E, Lucht L, Michael H, Beck JM, Curtis JL, Freeman CM, Morris A. Presence of Tropheryma whipplei in Different Body Sites in a Cohort of Healthy Subjects. Am J Respir Crit Care Med. 2016 Jul 15;194(2):243-5. doi: 10.1164/rccm.201601-0162LE. No abstract available. PMID 27420361
- [Derived] Dickson RP, Erb-Downward JR, Freeman CM, McCloskey L, Falkowski NR, Huffnagle GB, Curtis JL. Bacterial Topography of the Healthy Human Lower Respiratory Tract. mBio. 2017 Feb 14;8(1):e02287-16. doi: 10.1128/mBio.02287-16. PMID 28196961